CLINICAL TRIAL: NCT02176954
Title: The Influence of Adhesive Wafer Design on Fit to the Body
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: CP247
Record Dates: First submitted 2014-06-26; First posted 2014-06-27 (Estimated); Last update posted 2015-03-23 (Estimated); Status verified 2015-03

CONDITIONS: Ostomy - Ileostomy or Colostomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Test A, Test B, Comparator (Experimental): The subjects first test Coloplast Test A followed by Coloplast Test B and finally Comparator.
  Interventions: Device: Test A; Device: Test B; Device: Comparator
- Test A, Comparator, Test B (Experimental): The subjects first test Coloplast Test A followed by Comparator and finally Coloplast Test B.
  Interventions: Device: Test A; Device: Test B; Device: Comparator
- Test B, Test A, Comparator (Experimental): The subjects first test Coloplast Test B followed by Coloplast Test A and finally Comparator.
  Interventions: Device: Test A; Device: Test B; Device: Comparator
- Test B, Comparator, Test A (Experimental): The subjects first test Coloplast Test B followed by Comparator and finally Coloplast Test B.
  Interventions: Device: Test A; Device: Test B; Device: Comparator
- Comparator, Test A, Test B (Experimental): The subjects first test Comparator followed by Coloplast Test A and then Coloplast Test B
  Interventions: Device: Test A; Device: Test B; Device: Comparator
- Comparator, Test B, Test A (Experimental): The subjects first test Comparator followed by Coloplast Test B and then Coloplast Test A.
  Interventions: Device: Test A; Device: Test B; Device: Comparator

INTERVENTIONS:
Device: Test A — Test A is a new 1-piece ostomy appliance developed by Coloplast A/S
Device: Test B — Test B is a new 1-piece ostomy appliance developed by Coloplast A/S
Device: Comparator — Two comparators will be used: Moderma Flex (Hollister) or Confidence Natural drainable (Salts).These product are commercially available.
  Subjects will be randomized into one of twelwe arms. Data will be analyzed by pooling the two comparators, Moderma Flex and Confidence Natural, Drainable, why six arms are displayed.

SUMMARY:
The aim of this study is to investigate the influence of the adhesive wafer design on the products ability to fit to the body..

ELIGIBILITY:
Inclusion Criteria:

To participate in the study, it is mandatory that the subject fulfill all inclusions criteria:

* Have given written informed consent and signed letter of Authority
* Be at least 18 years of age and have full legal capacity
* Have had their ileostomy or colostomy for at least 3 months
* Have a stoma with a diameter between 15 and 43 mm
* Be able to handle the product themselves
* Be able to use a custom cut product
* Normally experience faeces under the adhesive wafer at least 3 times during 2 weeks
* Currently using a 1-piece flat product or a 1-piece soft convex product
* Be willing to test products with open bag size maxi
* Be willing to test Moderma Flex or Confidence® Natural, Drainable and the two test products A and B
* Be willing to use minimum 1 test product every second day, i.e. maximum 48 hours wear time per product
* Be suitable for participating in the investigation
* Be willing to take/have taken pictures of the stoma before, during and after application of product

Exclusion Criteria:

Subjects complying with the following criteria must be excluded from participation in the clinical investigation:

* Are currently receiving or have within the past 2 months received radio-and/or chemotherapy
* Are currently receiving or have within the past month received topical steroid treatment in the peri-stomal skin area or systemic steroid (tablet/injection) treatment
* Are pregnant or breastfeeding
* Are participating in other interventional clinical investigations or have previously participated in this investigation
* Use irrigation during the investigation (flush the intestines with water)
* Are currently suffering from peri-stomal skin problems i.e. bleeding and/or broken skin (assessed by the study nurse)
* Have a loop stoma
* Have known hypersensitivity towards any of the test products

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-07; Primary Completion 2015-02 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Fit to body | 14 +/- 2 days
  Subjects will evaluate the fit to body for each product by answering the question "How was the base plates ability to fit the body contours in the area around the stoma?"
  The question is answered with a 5-point scale ranging from Very Poor - Very Good (1-5), where the very poor (1) is the worst possible score and very good (5) is the best possible score.

CONTACTS AND LOCATIONS:
Overall Officials: Khalid Abd-Elaziz, MD, Principal Investigator — QPS Netherlands; Susanne Eyre, MD, Principal Investigator — Synexus North East, United Kingdom; Gillian Hopkins, Principal Investigator — Cheltenham General Hospital, United Kingdom
Locations (10):
- QPS Netherlands, Groningen, Netherlands
- United Kingdom (9):
  - Synexus Thames Valley, Berkshire
  - Synexus Midlands, Birmingham
  - Synexus Wales, Cardiff
  - Synexus Scotland, Glasgow
  - Cheltenham General Hospital, Gloucestershire
  - Synesxus Lancashire, Lancashire
  - Synexus Merseyside, Liverpool
  - Synexus Manchester, Manchester
  - Synexus North East, Northumberland